CLINICAL TRIAL: NCT06307197
Title: HAAL: HeAlthy Ageing Eco-system for peopLe With Dementia
Acronym: HAAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INRCA_008_2023
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-10

CONDITIONS: Dementia; Devices; Artificial Intelligence; Older People; Caregiver Burden
Keywords: dementia; caregiver; older people; technological devices; quality of life
MeSH Terms: conditions — Dementia; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- older adults (Experimental)
  Interventions: Device: HAAL platform

INTERVENTIONS:
Device: HAAL platform — The HAAL platform is composed by 6 devices (lifestyle monitoring system, a smart mattress, a GPS tracking system, a social robot, an interactive game for cognitive training, and an alarm system), 1 tablet and 1 dashboard. Each user benefits of a combination of such devices, according to its own needs. The dashboard, that is used by the Formal Caregiver, receives, analyses, and show data acquired by those devices.
  The platform uses Artificial Intelligence (AI) algorithms - in particular machine learning (ML) is used - to analyse the collected data. The main reason for using AI in HAAL is that the platform collects data from different sensors.

SUMMARY:
HAAL project aims to test several technological devices in order to improve the quality of life of older people with dementia and their informal and formal caregiver.

DETAILED DESCRIPTION:
The HAAL study is a feasibility study. The general objectives of the HAAL project is to be assessed the stress relief at work for formal and informal caregivers, the improvement in the perceived quality of life for informal caregivers and person with dementia, the reduction in case load for the formal caregivers and the increased cost-effectiveness of the HAAL solution in comparison to the available services. The experimentation will be carried out in 3 sites: Italy, The Netherlands and Taiwan. The study consists in a alpha phase (5 older adults with dementia, 5 formal caregivers and 5 formal caregivers) and in a beta phase (10 older adults with dementia, 10 formal caregivers and 10 formal caregivers).

ELIGIBILITY:
Inclusion Criteria:

* being the caregiver of a person with cognitive impairment or dementia;
* availability of time to participate;
* visit the assisted person at least two times at week or live with him/her.

Exclusion Criteria:

* Lack of written informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Care load of caregivers | baseline, 1, 2, and 3 months later
  The burden of the caregiver will be assessed through the ZARIT Burden Interview (ZBI). The ZBI is a caregiver self-report measure, containing 22 items. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always).Total score range: 0 to 88. score range 0-21: no to mild burden; score range 21-40: mild to moderate burden; score range 41-60: moderate to severe burden score ≥ 61: severe burden.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Bevilacqua, Study Director — IRCCS INRCA
Locations (1):
- IRCCS INRCA Hospital, Ancona, Italy